CLINICAL TRIAL: NCT03853785
Title: The Efficacy of Intralesional Measles, Mumps, Rubella (MMR) Vaccine, Intralesional Candidal Antigen and Topical Podophyllin in Treatment of Genital Warts: A Comparative Study
Brief Title: Efficacy of Intralesional MMR Vaccine,Intralesional Candidal Antigen&Topical Podophyllin in Treatment of Genital Warts
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Meriam Mamdouh Boshra, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MMR vaccine in genital warts
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Condylomata Acuminata
MeSH Terms: conditions — Condylomata Acuminata | interventions — Measles-Mumps-Rubella Vaccine; PRA1 protein, Candida albicans; Podophyllin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intralesional MMR vaccine (Active Comparator): Intralesional Mumps, measles and rubella (MMR) vaccine in genital warts
  Interventions: Biological: MMR vaccine
- intralesional candida antigen (Active Comparator): intralesional candida antigen in genital warts
  Interventions: Biological: Candida antigen
- Topical Podophyllin (Active Comparator): Topical Podophyllin in genital warts
  Interventions: Drug: Topical Podophyllin

INTERVENTIONS:
Biological: MMR vaccine — Intralesional injection of 0.5 ml MMR vaccine in the largest lesion . Injections will be repeated into the same lesion every 2 weeks for a maximum of three treatment sessions.
  Arms: Intralesional MMR vaccine
Biological: Candida antigen — Intralesional injection of Candidal antigen with a dose of (0.1ml -0.3ml) by an insulin syringe in the largest wart at the first visit. Injections will be repeated for all patients into the same lesion every 2 weeks for a maximum of three treatment sessions.
  Arms: intralesional candida antigen
Drug: Topical Podophyllin — It will be applied to the wart by using a cotton tipped swab once a week . The procedure will be limited to 10 cm2 per session .Surrounding skin will be protected by Vaseline. Podophyllin will be washed 4 hour after application . The procedure will be repeated every week till 6 weeks .
  Arms: Topical Podophyllin

SUMMARY:
This study compares the safety and efficacy of intralesional Candidal antigen versus Intralesional MMR vaccine versus podophyllin for treatment of genital warts.

DETAILED DESCRIPTION:
Anogenital human papillomavirus (HPV) is a highly prevalent sexually transmitted infection ,seen predominantly in young adults.

Condyloma acuminata or benign anogenital warts are typically caused by HPV-6 OR 11 which are considered low risk types.Persistent infection with high risk HPV types predominantly HPV-16 and 18 is the primary and major cause of cervical cancers and a subset of vaginal,vulvar, penile , anal ,oropharyngeal and rarely squamous cell carcinoma of the digits.

Warts may reflect a localized or systemic cell-mediated immune (CMI) deficiency to HPV.

Anogenital warts may appear as a single lesion or in clusters as flat, flesh-coloured to pigmented plaques or rough-surfaced papules and exophytic nodules.

The conventional modalities in treatment of warts include destructive therapies such as salicylic acid, trichloroacetic acid, cryotherapy, silver nitrate, phenol, cantharidin, surgical interventions and lasers; antiproliferative agents such as bleomycin, podophyllin, podophyllotoxin, and 5-fluro uracil; antiviral agents such as cidofovir and retinoids.

Because of the cumbersome nature of these procedures and a high risk of recurrence, immunotherapy is becoming more and more popular, especially in the treatment of refractory cutaneous and genital warts.It enhances recognition of the virus by the immune system. immunotherapy not only causes a resolution of the treated wart but also leads to clearance of distant warts, at least in a subset of the responders.

Immunotherapy in warts can be administered by various methods. The first method is topical application of certain inorganic molecules that are capable of eliciting a contact hypersensitivity reaction with secondary activation of an immunological response .or even topical applications of immune modulators like imiquimod,A second modality is the use of oral immune modulators such as cimetidine,and levamisole .

A third method is Intralesional injection of immunotherapeutic agent that utilizes the ability of the immune system to mount a delayed type hypersensitivity response to various antigens and also the wart tissue leading to production of Th1 cytokines which activate cytotoxic and natural killer cells to eradicate HPV infection.

Immunotherapy with different skin test antigens like Candida, mumps or trichophyton antigen is a relatively new treatment option for warts. Candida antigen reported success in majority of patients treated with this test antigen .

Mumps, measles and rubella (MMR) vaccine is a freeze-dried preparation of live attenuated strains of measles, mumps and rubella viruses (0.5 ml/dose). In some of the previous studies, it has been shown that mumps-measles-rubella (MMR) vaccine results in regression of warts via immunomodulation and induction of immune system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with anogenital warts with ages ranging from 3 to 50 years
* Genital warts resistant to treatment
* Genital warts that had relapsed at least once after treatment with any of the tissue-destructive modalities.

Exclusion Criteria:

* Patients with any evidence of immunosuppression
* Eczematous skin disorder
* Those with any history of hypersensitivity to Candida albicans antigen
* Pregnant or lactating women.

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Cure rate | 45 days
  Assess cure rate of MMR vaccine and candida antigen and topical podophyllin in treatment of genital warts (complete disappearance of lesions) in 45 days duration and compare efficacy of the measures.